CLINICAL TRIAL: NCT05496764
Title: The Therapeutic Effect and Quality of Life After Local Injection of Steroid VS. Glucose 5% for Carpal Tunnel Syndrome : Double-blinded Clinical Trial
Brief Title: Local Injection of Steroid VS.Glucose 5% in Carpal Tunnel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Talaat Helmy Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22151125
Record Dates: First submitted 2021-12-27; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: local injection; pain relief; steroid; glucose 5%
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Dexamethasone; Glucose

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The patients were randomly assigned to one of two groups. Serially numbered opaque closed envelopes were used for allocation concealment. Allocation was maintained. To ensure double blinding, the random allocation sequence was kept by one investigator different from the one who enrolled the participants or assigned them to the interventions. Moreover, a third investigator was responsible for following the patients up and for assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): 26 patients we planned to inject them local steroid( 4 mg of dexamethasone acetate combined with 1% lidocaine into the carpal tunnels) directly into the carpal tunnel in (group A)
  Interventions: Drug: Dexamethasone; Drug: Glucose Injection
- Group B (Active Comparator): 26 patients we planned to inject them local glucose 5% ( 10 ml glucose) directly into the carpal tunnel in (group A)
  Interventions: Drug: Dexamethasone; Drug: Glucose Injection

INTERVENTIONS:
Drug: Dexamethasone — we planned to inject steroid( 4 mg of dexamethasone acetate combined with 1% lidocaine into the carpal tunnels) directly into the carpal tunnel in group A
Drug: Glucose Injection — inject10 ml glucose 5% into the carpal tunnel in group B
  Other Names: glucose 5%

SUMMARY:
To assess pain relief and quality of life among patients with carpal tunnel syndrome after local steroid vs. glucose 5% injection.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most prevalent type of peripheral nerve entrapment involving compression of the median nerve in the carpal tunnel. 1 This condition is more common in females than in males. CTS may be unilateral or bilateral. It is a significant cause of morbidity and poor quality of life in those patients. There is deterioration in functional outcomes and maybe psychologically as well. The severity of CTS varied from mild to moderate to severe. Its signs and symptoms include numbness along with the median nerve distribution of the hand, pain, atrophy of muscles, handgrip weakness, etc. Mild or moderate cases are usually seeking conservative treatment like electrotherapeutic modalities, manual therapy interventions, oral supplements and medications, and wrist immobilizations such as splints. Severe cases are likely to go toward surgery. But most patients with CTS are reluctant to take the surgical choice, mainly because of financial issues and secondary complications. Therefore, the evaluation of the effectiveness of the non-surgical (conservative) therapies should be a major concern, as they are cost-effective and lacks secondary complications. Much research has been conducted to see the efficacy of various conservative therapies.

-study method: We are going to carry out a double-blinded randomized, case-controlled study on 52 patients who are randomly chosen and categorized them into 2 groups, 26 patients each. we planned to inject steroid( 4 mg of dexamethasone acetate combined with 1% lidocaine into the carpal tunnels) directly into the carpal tunnel in (group 1) and to inject 10 ml glucose 5% into the carpal tunnel for the other group (group 2).. All injections will be under sonographic guidance. Neurophysiology, U/S, pain scales, and quality of life scales studies will be performed for these two groups before treatment and after 12 weeks of injection. The patients will be followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. female or male patient > 18y
2. mild to moderate cases of carpal tunnel syndrome according to Bland's Neurophysiological Grading Scale for Patients with CTS
3. clear consent to participate in the study

Exclusion Criteria:

1. age younger than 18y.
2. severe cases of CTS.
3. systemic diseases cause CTS .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
the changes in visual analogue scale (pre - post- and follow up) | 14 days
  the changes in visual analogue scale (pre - post- and follow up) Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores . pain intensity described as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
-To evaluate the effect of sonar guided steroid vs. glucose 5% injection on U/S (pre-post and follow up). | 3 months
  To evaluate the effect of sonar guided steroid vs. glucose 5% injection on U/S (pre-post and follow up).
  -U/S In the literature, four criteria are used to diagnose CTS by sonography:
  1. Increase in cross-sectional area at the level of the pisiform bone;
  2. Increase in the flattening ratio at the level of the hook of the Hamate
  3. Palmar bowing of the flexor retinaculum by sonography.
  The above readings will be calculated and will be compared to the previous readings of the same patient of each group.
  eg. The grade of CTS severity was classified according to the CSA of the median nerve considering 10.0 - 12.9mm2 as mild grade, 13.0 - 15.0mm2 as moderate grade and >15.0 mm2 as severe grade
To evaluate the effect of sonar guided steroid vs. glucose 5% injection on neurophysiological studies (pre-post and follow up). | 3 months
  To evaluate the effect of sonar guided steroid vs. glucose 5% injection on neurophysiological studies (pre-post and follow up).
  Neurophysiology studies (sensory, motor conduction, and f wave of both median and ulnar nerve)
  Grade ............................................ EDX Abnormality
  1. Very mild CTS ............ .................. detected by only PWDSLD*
  2. Mild Median.................................... DML <4.5 and sensory NCV <40
  3. Moderately severe Median............. DML♦ >4.5 and <6.5 with preserved SNAP
  4. Severe Median ...............................DML >4.5 and <6.5 with absent SNAP
  5. Very severe Median....................... DML >6.5 with CMAP >0.2 mv
  6. Extremely severe Median ...............CMAP from APB <0.2 mv
  we detect improvment in latency, amplitude and NCV after 3 months of local injection and comparing it with previous readings of the same patient of each group.

CONTACTS AND LOCATIONS:
Overall Officials: Eman MH Khedr, Study Director — Assiut University; Khaled O Aboshaera, Study Director — Assiut University; Aml MA Tohami, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Wipperman J, Goerl K. Carpal Tunnel Syndrome: Diagnosis and Management. Am Fam Physician. 2016 Dec 15;94(12):993-999. PMID 28075090
- [Background] Kamel SR, Sadek HA, Hamed A, Sayed OA, Mahmud MH, Mohamed FA, El Sagher GM, Aly LH. Ultrasound-guided insulin injection for carpal tunnel syndrome in type 2 diabetes mellitus patients. Clin Rheumatol. 2019 Oct;38(10):2933-2940. doi: 10.1007/s10067-019-04638-7. Epub 2019 Jun 17. PMID 31209710
- [Background] Ashraf A, Moghtaderi AR, Yazdani AH, Mirshams S. Evaluation of effectiveness of local insulin injection in non-insulin-dependent diabetic patient with carpal tunnel syndrome. Electromyogr Clin Neurophysiol. 2009 May-Jun;49(4):161-6. PMID 19534294
- [Background] Pourmemari MH, Shiri R. Diabetes as a risk factor for carpal tunnel syndrome: a systematic review and meta-analysis. Diabet Med. 2016 Jan;33(1):10-6. doi: 10.1111/dme.12855. Epub 2015 Aug 18. PMID 26173490
- [Background] Nakandala, Piumi. (2019). International Journal of Advanced Research and Publications Manual Therapy Interventions For Carpal Tunnel Syndrome: A Review. 3. 88-96.
- [Background] Recio-Pinto E, Rechler MM, Ishii DN. Effects of insulin, insulin-like growth factor-II, and nerve growth factor on neurite formation and survival in cultured sympathetic and sensory neurons. J Neurosci. 1986 May;6(5):1211-9. doi: 10.1523/JNEUROSCI.06-05-01211.1986. PMID 3519887
- [Background] Kanikannan MA, Boddu DB, Umamahesh, Sarva S, Durga P, Borgohain R. Comparison of high-resolution sonography and electrophysiology in the diagnosis of carpal tunnel syndrome. Ann Indian Acad Neurol. 2015 Apr-Jun;18(2):219-25. doi: 10.4103/0972-2327.150590. PMID 26019423
- [Background] Mody GN, Anderson GA, Thomas BP, Pallapati SC, Santoshi JA, Antonisamy B. Carpal tunnel syndrome in Indian patients: use of modified questionnaires for assessment. J Hand Surg Eur Vol. 2009 Oct;34(5):671-8. doi: 10.1177/1753193409101469. Epub 2009 Aug 17. PMID 19687086
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Arian M, Mirmohammadkhani M, Ghorbani R, Soleimani M. Health-related quality of life (HRQoL) in beta-thalassemia major (beta-TM) patients assessed by 36-item short form health survey (SF-36): a meta-analysis. Qual Life Res. 2019 Feb;28(2):321-334. doi: 10.1007/s11136-018-1986-1. Epub 2018 Sep 7. PMID 30194626
- [Background] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Sharour LA, Omari OA, Salameh AB, Yehia D. Health-related quality of life among patients with colorectal cancer. J Res Nurs. 2020 Mar;25(2):114-125. doi: 10.1177/1744987119846177. Epub 2019 Aug 22. PMID 34394615
- [Background] Wong SM, Griffith JF, Hui AC, Lo SK, Fu M, Wong KS. Carpal tunnel syndrome: diagnostic usefulness of sonography. Radiology. 2004 Jul;232(1):93-9. doi: 10.1148/radiol.2321030071. Epub 2004 May 20. PMID 15155897
- [Background] Kele H, Verheggen R, Bittermann HJ, Reimers CD. The potential value of ultrasonography in the evaluation of carpal tunnel syndrome. Neurology. 2003 Aug 12;61(3):389-91. doi: 10.1212/01.wnl.0000073101.04845.22. PMID 12913205
- [Background] Bland JD. A neurophysiological grading scale for carpal tunnel syndrome. Muscle Nerve. 2000 Aug;23(8):1280-3. doi: 10.1002/1097-4598(200008)23:83.0.co;2-y. PMID 10918269
- [Background] Subandi, S., Mirawati, D., Erdana Putra, S., Hafizhan, M., Susilo, W. and Danuaji, R., 2020. THE RELATIONSHIP BETWEEN WORKING PERIOD OF BATIK CRAFTSMEN AND INCIDENT OF CARPAL TUNNEL SYNDROME. MNJ (Malang Neurology Journal), 6(2), pp.73-76
- [Background] Ezzati K, Laakso EL, Saberi A, Yousefzadeh Chabok S, Nasiri E, Bakhshayesh Eghbali B. A comparative study of the dose-dependent effects of low level and high intensity photobiomodulation (laser) therapy on pain and electrophysiological parameters in patients with carpal tunnel syndrome. Eur J Phys Rehabil Med. 2020 Dec;56(6):733-740. doi: 10.23736/S1973-9087.19.05835-0. Epub 2019 Nov 18. PMID 31742366
- [Background] Maeda Y, Kim H, Kettner N, Kim J, Cina S, Malatesta C, Gerber J, McManus C, Ong-Sutherland R, Mezzacappa P, Libby A, Mawla I, Morse LR, Kaptchuk TJ, Audette J, Napadow V. Rewiring the primary somatosensory cortex in carpal tunnel syndrome with acupuncture. Brain. 2017 Apr 1;140(4):914-927. doi: 10.1093/brain/awx015. PMID 28334999
- [Background] Niempoog S, Sanguanjit P, Waitayawinyu T, Angthong C. Local injection of dexamethasone for the treatment of carpal tunnel syndrome in pregnancy. J Med Assoc Thai. 2007 Dec;90(12):2669-76. PMID 18386719
- [Background] Sung YT, Wu JS. The Visual Analogue Scale for Rating, Ranking and Paired-Comparison (VAS-RRP): A new technique for psychological measurement. Behav Res Methods. 2018 Aug;50(4):1694-1715. doi: 10.3758/s13428-018-1041-8. PMID 29667082